CLINICAL TRIAL: NCT05771870
Title: Pediatric Nursing Students' Self-efficacy Regarding Pediatric Medication Administration and, Clinical Comfort and Worry: a Study on a Two-group Pre-post-test Design Comparing Nurse and Peer Mentoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Özlem Öztürk Şahin, Associate professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KBU-OOSahin-001
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Medication Administration; Mentoring; Comfort
Keywords: medication administration; mentoring; nursing students

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer mentoring (Experimental): The clinical practice day of the Child Health and Diseases Nursing course included mentoring practice. This is a 3rd-grade (5th semester) course that includes 6 hours of theory and 8 hours of practice in the applicable curriculum. The clinical practice of the Child Health and Diseases Nursing course is carried out for 14 weeks (one semester) 1 day a week at the Children's Units of the Karabük Training and Research Hospital in the program in which the study was done. Throughout all clinical practice days, mentors chosen from graduate students followed the students in the peer mentorship group during the medication preparation and administration processes, providing feedback on their positive, negative, or inadequacies.
  Interventions: Other: Peer mentoring
- Nurse mentoring (Experimental): The clinical practice day of the Child Health and Diseases Nursing course included mentoring practice. This is a 3rd-grade (5th semester) course that includes 6 hours of theory and 8 hours of practice in the applicable curriculum. The clinical practice of the Child Health and Diseases Nursing course is carried out for 14 weeks (one semester) 1 day a week at the Children's Units of the Karabük Training and Research Hospital in the program in which the study was done. Mentors from the clinical nursing community attended the students in the nurse mentoring group during the drug preparation and administration processes and provided feedback on their positive, negative, or inadequacies.
  Interventions: Other: Nurse mentoring

INTERVENTIONS:
Other: Peer mentoring — Mentoring is a support network in which a more talented or experienced individual serves as a role model for a less talented individual in order to encourage professional and personal growth. Mentoring improves students' learning, abilities, and self-efficacy while decreasing stress and anxiety in nursing students through more effective communication, collaborative learning, and critical thinking.
  After understanding about the study, two master's degree students from Karabük University Institute of Graduate Studies of Child Health and Diseases Nursing consented to participate on a volunteer basis and became peer mentors in the study. All postgraduate students are pediatric nurses with at least two years of clinical experience who have completed their undergraduate nursing program.
  Arms: Peer mentoring
Other: Nurse mentoring — Mentoring is a support network in which a more talented or experienced individual serves as a role model for a less talented individual in order to encourage professional and personal growth. Mentoring improves students' learning, abilities, and self-efficacy while decreasing stress and anxiety in nursing students through more effective communication, collaborative learning, and critical thinking.
  After providing information about the research to bachelor's degree nurses who have worked in the Children's Units of Karabuk Training and Research Hospital for at least two years, two mentors for the nurse mentoring group were chosen on a volunteer basis. Mentors were taught on the concept of mentoring, the roles of the mentor, interpersonal relationships, and communication skills prior to the study.
  Arms: Nurse mentoring

SUMMARY:
Children are a particularly vulnerable population to medication mistakes, and it is critical to improve the self-efficacy, clinical comfort, and worry levels of student nurses who will care with them. As a result, the purpose of this study was to investigate the effects of postgraduate nursing students' and clinical nurses' mentoring practice on pediatric nursing students' self-efficacy in pediatric medication administration, clinical comfort, and worry levels. The nurse mentoring group finished the study with 70 students, while the peer mentoring group (postgraduate nursing students) completed the study with 73 students, for a total of 143 students. For data collection, the "Participant Information Form," the "Medication Administration Self-Efficacy Scale in Children for Nursing Students," and the "Pediatric Nursing Students Clinical Comfort and Worry Tool" were utilized. The data is still being analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Third-year student at Department of Nursing
* Taking a Child Health and Disease Nursing course
* Successful completion of the Pharmacology course in the first year (2nd semester)
* Participating in research as a volunteer

Exclusion Criteria:

- Failure in the pharmacology course

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Change from medication administration self-efficacy scale in children for nursing students mean score at one semester (14 weeks). | Medication Administration Self-Efficacy Scale in Children for Nursing Students was used before the mentoring practice and when the mentoring practice ended (14 weeks later).
  This scale assesses nursing students' self-efficacy in medication preparation and administration for pediatric patients. The scale yields a lowest score of 16 and a top score of 80. The higher the score, the greater the students' sense of self-efficacy in pediatric medication administration.
Change from pediatric nursing students' clinical comfort and worry tool mean score at one semester (14 weeks). | Pediatric Nursing Students Clinical Comfort and Worry Tool was used before the mentoring practice and when the mentoring practice ended (14 weeks later).
  This scale is used to assess nursing students' feelings of worry and comfort while working in pediatric clinics. The clinical comfort sub-dimension receives the lowest 6 and greatest 24 scores. The worry sub-dimension receives the lowest 5 and maximum 20 scores. Greater degrees of comfort and worry are indicated by higher scores on the comfort and worry parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabuk training and research hospital, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No